CLINICAL TRIAL: NCT06663293
Title: Comparison of High Flow and Conventional Nasal Cannula Outcomes in Pediatric Burn Patients Under Sedoanalgesia: A Prospective Randomized Study
Brief Title: Comparison of High Flow vs Standard Nasal Cannula in Children With Burns Under Sedoanalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeliha Alicikus (Other Government)
Responsible Party: Sponsor-Investigator, Zeliha Alicikus, Study Director, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01-93
Record Dates: First submitted 2024-10-17; First posted 2024-10-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Burns
Keywords: Pediatrics; Burn; Sedo-analgesia; Oxygen therapy; High flow Nasal Oxygen; Hypoxia
MeSH Terms: conditions — Burns; Hypoxia | interventions — Midazolam; Ketamine; Propofol

STUDY DESIGN:
Intervention Model Description: 50 patients aged 1-14 years in the pediatric burn unit were divided into two groups as Group HFO: High flow oxygen (n: 25) and Group NC: nasal cannula oxygen (n: 25).
  The high flow group received nasal high flow therapy delivered by AIRVO™ 2 (Fisher and Paykel Healthcare Systems, New Zealand) along with single-use nasal oxygen cannulas. The HFNCO device was set to a temperature of 36°C and an FiO2 of 0.4. The initial oxygen flow rate for the high flow group was determined according to the age and weight of the patients, based on our pediatric intensive care team's guidelines and the reference from the Slain NK (10) study. When SpO2 fell below 94%, it was considered hypoxia, and the flow rate was increased by 2 to 4 L/min.
  For the low flow group, the initial flow rate for nasal cannula oxygen was set at 3 L/min. In cases of hypoxia, the oxygen concentration was adjusted by increasing the flow rate by 1 to 2 L/min.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Nasal Cannula Oxygen group (Placebo Comparator): Participants received low flow oxygen therapy through a conventional nasal cannula. The initial flow rate for nasal cannula oxygen was set at 3 L/min. In cases of hypoxia, the oxygen concentration was adjusted by increasing the flow rate by 1 to 2 L/min.
  Interventions: Other: Conventional Nasal Cannula; Drug: midazolam, ketamine, propofol; Drug: Propofol
- High-flow Nasal Cannula Oxygen Group (Active Comparator): Participants received nasal high flow therapy delivered by AIRVO™ 2 (Fisher and Paykel Healthcare Systems, New Zealand) along with single-use nasal oxygen cannulas.
  Interventions: Other: High-flow nasal cannula; Drug: midazolam, ketamine, propofol; Drug: Propofol

INTERVENTIONS:
Other: Conventional Nasal Cannula — The initial flow rate for nasal cannula oxygen was set at 3 L/min. In cases of hypoxia, the oxygen concentration was adjusted by increasing the flow rate by 1 to 2 L/min.
  Arms: Conventional Nasal Cannula Oxygen group
Other: High-flow nasal cannula — The high-flow nasal oxygenation device was set to a temperature of 36°C and an FiO2 of 0.4. The initial oxygen flow rate for the high flow group was determined according to the age and weight of the patients, based on our pediatric intensive care team's guidelines and the reference from the Slain study. When SpO2 fell below 94%, it was considered hypoxia, and the flow rate was increased by 2 to 4 L/min.
  Arms: High-flow Nasal Cannula Oxygen Group
Drug: midazolam, ketamine, propofol — Sedation was done with IV midazolam 0.025 to 0.1 mg/kg, IV ketamine 0.25 to 0.5 mg/kg, and IV propofol (1%) 0.25 to 0.5 mg/kg
Drug: Propofol — Sedation maintenance was done by propofol 0.5 to 1 mg/kg/h

SUMMARY:
The aim of this study is to investigate the positive effects of high-flow oxygen therapy on the reduction of airway adverse events and recovery time compared to conventional nasal oxygen therapy in pediatric burns treated with procedural sedoanalgesia.

DETAILED DESCRIPTION:
High flow nasal cannula oxygenation (HFNCO) has gained popularity in pediatric anesthesia practice. The basic mechanism of HFNCO involves reducing metabolic cost and work of breathing, decreasing nasopharyngeal resistance, and improving gas conditioning and secretion clearance. Heating and humidifying the oxygen administered make it easier for patients to tolerate high flow. The flow rate can be adjusted for all age groups. However, there are no studies in the literature investigating the effectiveness of HFNCO during procedural sedation in pediatric burn patients.

This randomized prospective study was performed in 50 patients aged 1-14 years in the pediatric burn unit. Patients were divided into two groups as Group HFO: High flow oxygen (n: 25) and Group NC: nasal cannula oxygen (n: 25). Age, sex, burn percentage, concomitant diseases, ASA score, BMI (body mass index), respiratory and hemodynamic parameters, recovery time and presence of complications during sedoanalgesia were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age: 1 and 14 years
* ASA risk groups 1-3
* Second-degree burns covering more than 10% of the total body surface area, or third- and fourth-degree burns covering more than 2% of the total body surface area, burns involving the face, hands, feet, genital area, perineum, or major joints, electrical burns, and chemical burns.

Exclusion Criteria:

* Under 1 year of age or over 14 years of age
* ASA score above 3
* Having restrictive or obstructive chronic respiratory diseases, active upper or lower respiratory infections, first-degree burns, and burns to the nasal area or respiratory tract.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Heart rate in beats per minute | Intraoperative measurements will be taken at 0, 5, 15, 20 minutes and Postoperative measurements will be taken at 0, 5, and 10 minutes
  Heart rate in beats per minute using ECG leads will be measured intraoperatively and postoperatively
Respiratory rate in breaths per minute | Intraoperative measurements will be taken at 0, 5, 15, 20 minutes and Postoperative measurements will be taken at 0, 5, and 10 minutes
  Respiratory rate in breaths per minute will be measured intraoperatively and post-operatively
SpO2 in percentage | Intraoperative measurements will be taken at 0, 5, 15, 20 minutes and Postoperative measurements will be taken at 0, 5, and 10 minutes
  SpO2 in percentage will be measured intraoperatively and post-operatively
End-tidal CO2 in mmHg | Intraoperative measurements will be taken at 0, 5, 15, 20 minutes and Postoperative measurements will be taken at 0, 5, 10 minutes and at recovery time60 minutes
  End-tidal CO2 in mmHg will be measured intraoperatively and post-operatively
Oxygen flow levels in Liters per minute | Intraoperative measurements will be taken at 0, 5, 15, 20 minutes
  Oxygen flow levels in Liters per minute will be measured intraoperatively

SECONDARY OUTCOMES:
Need for oxygen assessed by SpO2 | Intraoperative measurements will be taken at 0, 5, 15, 20 minutes and Postoperative measurements will be taken at 0, 5, and 10 minutes
  Need for oxygen assessed by SpO2 measured in percentage intraoperatively and post-operatively. SpO2 <94% is considered desaturation
Need for oxygen assessed by Near-Infrared Spectroscopy (NIRS) | Intraoperative measurements will be taken at 0, 5, 15, 20 minutes
  Need for oxygen assessed by Near-Infrared Spectroscopy (NIRS) measured intraoperatively. 20% drop from the individual's baseline will be considered desaturation

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No